CLINICAL TRIAL: NCT03692403
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Trial Assessing the Efficacy, Safety and Dose-response of Quinagolide Extended-release Vaginal Rings Administered Sequentially for 4 Menstrual Cycles in Women With Moderate to Severe Endometriosis-related Pain
Brief Title: Randomized Trial Assessing Quinagolide Vaginal Ring for Endometriosis-related Pain
Acronym: RAQUEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000165
Record Dates: First submitted 2018-09-14; First posted 2018-10-02 (Actual); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2022-10

CONDITIONS: Endometriosis-related Pain
MeSH Terms: interventions — quinagolide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Quinagolide 360 µg (Experimental): Vaginal ring containing Quinagolide 360 μg, with daily target release rate of 4.5 μg
  Interventions: Drug: Quinagolide 360 µg
- Quinagolide 720 µg (Experimental): Vaginal ring containing Quinagolide 720 μg, with daily target release rate of 9 μg
  Interventions: Drug: Quinagolide 720 µg
- Quinagolide 1080 µg (Experimental): Vaginal ring containing Quinagolide 1080 μg, with daily target release rate of 13.5 μg
  Interventions: Drug: Quinagolide 1080 µg
- Placebo (Placebo Comparator): Vaginal ring containing matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quinagolide 360 µg — Vaginal ring containing quinagolide 360 µg for daily releases
  Other Names: FE 999051
  Arms: Quinagolide 360 µg
Drug: Quinagolide 720 µg — Vaginal ring containing quinagolide 720 µg for daily releases
  Other Names: FE 999051
  Arms: Quinagolide 720 µg
Drug: Quinagolide 1080 µg — Vaginal ring containing quinagolide 1080 µg for daily releases
  Other Names: FE 999051
  Arms: Quinagolide 1080 µg
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of three doses of quinagolide administered as an extended-release vaginal ring compared to placebo on reduction of moderate to severe endometriosis-related pain

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal females aged ≥18 years at time of signing informed consent(s) with regular menstrual cycles.
* Body mass index (BMI) of 18-42 kg/m2 (both inclusive) at screening.
* Initial confirmation of endometriosis by laparoscopy or laparotomy within the last 10 years before the run-in visit or visualization of persistent endometrioma by repeat ultrasound.
* Transvaginal ultrasound documenting a uterus with no clinically significant abnormalities and presence of at least one ovary with no clinically significant abnormalities (with the exception of endometrioma) at the run-in visit.
* Eligible participants experienced moderate to severe endometriosis-related pain, which was defined as at the run-in visit, the participant having an NRS score of ≥5 for the worst endometriosis related pain during the past menstrual cycle and at randomization, the participant having a mean daily NRS score of ≥4 for the worst endometriosis related pain during each run-in menstrual cycle.

Exclusion Criteria:

* History of no relief of endometriosis related pain after any medical therapy or surgery. However, history of partial pain relief, discontinuation due to side effects are not exclusionary.
* Known bone diseases (e.g. osteoporosis, Paget's disease and osteomalacia) affecting bone resorption or bone formation markers.
* Any significant abnormal findings of heart examinations before randomization.
* History of mental illness including occurrence of acute psychosis, bipolar disorders and schizophrenia (except for well-controlled anxiety and/or depression with no changes to interventions for 6 months prior to start of run-in)
* History of impulse control disorders including pathological gambling, compulsive buying, hypersexuality, and binge eating or being identified with potential impulse control disorder by the questionnaire for impulsive-compulsive disorders (a score ≥2 for any sub-questions of Question 3 or a score ≥1 for any sub-questions of Question 4) prior to randomization.
* History of orthostatic hypotension or recurrent syncope.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (43):
- United States (43):
  - Marchand Institute for Minimally Invasive Surgery, Mesa, Arizona
  - Arkansas Primary Care Clinic, Little Rock, Arkansas
  - Medical Center for Clinical Research, San Diego, California
  - UConn Health Lowell P Weicker Jr Clinical Research Center, Farmington, Connecticut
  - Yale Fertility Center, New Haven, Connecticut
  - Omega Research Consultants, DeBary, Florida
  - South Florida Research Center, Miami, Florida
  - Florida Research Center, Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Vista Health Research, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Physician Care Clinical Research, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Advance Clinical Research, Meridian, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - The Iowa Clinic, Ankeny, Iowa
  - Cypress Medical Research Center, Wichita, Kansas
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Omni Fertility Clinical Research LLC, Shreveport, Louisiana
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - OB/Gyn Associates, Silver Spring, Maryland
  - Onyx Clinical Research, Flint, Michigan
  - Valley OB/GYN Clinic, PC, Saginaw, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - OB•GYN Associates of WNY, West Seneca, New York
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Carolina's Women's Research and Wellness Center, Durham, North Carolina
  - Rapha Institute For Clinical Research, Fayetteville, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Unified Women's Clinical Research d/b/a Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Main Line Fertility Center, Bryn Mawr, Pennsylvania
  - Penn State Health - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Austin Area Ob, Gyn and Fertility, Austin, Texas
  - Corpus Christi Women's Clinic, Corpus Christi, Texas
  - Advances in Health, Inc., Houston, Texas
  - Center of Reproductive Medicine LLC, Webster, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Tidewater Clinical Research, Inc., Norfolk, Virginia
  - OB/GYN Specialists of Richmond, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed in 12 investigational sites in the US between Dec 2018 and Feb 2022
Pre-assignment Details: In total, 107 participants were screened. Of these, 85 were screening failures and 22 were randomized. All the randomized participants were exposed to the investigational medical product (IMP): 6 participants to Quinagolide 360 µg, 5 participants to Quinagolide 720 µg, 8 participants to Quinagolide 1080 µg and 3 participants to Placebo.
Period: Overall Study
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Started | 6 | 5 | 8 | 3
Completed | 5 | 4 | 6 | 2
Not Completed | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 8 | 3 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 8 | 3 | 22
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (8.22) | 33.2 (9.36) | 37.5 (6.65) | 32.0 (5.20) | 33.6 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 8 | 3 | 22
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 0 | 5
  Not Hispanic or Latino | 5 | 3 | 6 | 3 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 1 | 4
  White | 6 | 4 | 6 | 2 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 8 | 3 | 22
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.33 (5.428) | 26.58 (5.006) | 29.91 (5.038) | 32.33 (7.190) | 29.05 (5.348)
Numerical Rating Scale (NRS) at baseline [Number; unit: Participants] — At baseline this is the numerical rating scale (NRS) for the worst endometriosis-related pain. The NRS is an 11-point scale, with 0 indicating no pain and 10 indicating the worst imaginable pain. Higher values represent a worse outcome.
  Participants
    6 | 1 | 0 | 0 | 0 | 1
    7 | 0 | 1 | 2 | 0 | 3
    8 | 2 | 1 | 1 | 0 | 4
    9 | 2 | 2 | 4 | 2 | 10
    10 | 1 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Mean Daily Numerical Rating Scale (NRS) Scores for the Worst Endometriosis-related Pain.
Description: Assessed daily by participants in an e-Diary. NRS is an 11-point scale, with 0 indicating no pain and 10 indicating the worst imaginable pain.
  Changes from baseline to cycle 4.
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 3 | 6 | 2
score on a scale | -0.66 (1.213) | -2.04 (2.092) | -2.14 (1.344) | -3.68 (1.685)

2. Secondary Outcome: Changes in the Mean Daily Numerical Rating Scale (NRS) Scores for the Worst Endometriosis-related Pain on Days With Menstrual Bleeding and for the Worst Endometriosis-related Pain on Days With no Menstrual Bleeding
Description: Assessed daily by participants in an e-Diary. NRS is an 11-point scale, with 0 indicating no pain and 10 indicating the worst imaginable pain.
  Days with menstrual bleeding (dysmenorrhea). No menstrual bleeding (non-menstrual pelvic pain) Changes from baseline to cycle 4
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 4 | 6 | 2
score on a scale
  Dysmenorrhea | -0.51 (0.989) | -3.70 (3.252) | -2.54 (1.787) | -4.90 (0.495)
  Non-menstrual pelvic pain | -0.69 (1.236) | -2.04 (2.390) | -2.08 (1.274) | -3.37 (2.040)

3. Secondary Outcome: Changes in the Mean Daily Numerical Rating Scale (NRS) Scores for the Worst Endometriosis-related Pain.
Description: Assessed daily by participants in an e-Diary. NRS is an 11-point scale, with 0 indicating no pain and 10 indicating the worst imaginable pain.
  Changes over 4 menstrual cycles
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 7 | 2
score on a scale
  Cycle 1 | -0.33 (1.200) | -1.42 (0.990) | -0.51 (0.733) | -1.97 (1.397)
  Cycle 2 | -0.79 (1.343) | -2.39 (3.127) | -1.63 (1.254) | -1.16 (1.190)
  Cycle 3: number analyzed (Participants) | 5 | 4 | 6 | 2
  Cycle 3 | -0.61 (1.057) | -1.71 (1.788) | -1.51 (1.912) | -2.29 (2.152)
  Cycle 4: number analyzed (Participants) | 5 | 3 | 6 | 2
  Cycle 4 | -0.66 (1.213) | -2.04 (2.092) | -2.14 (1.344) | -3.68 (1.685)

4. Secondary Outcome: Changes in the Mean Daily Numerical Rating Scale (NRS) Scores for the Worst Dysmenorrhea.
Description: as for outcome 3
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 7 | 2
score on a scale
  Cycle 1 | -1.10 (1.051) | -1.48 (1.690) | -0.61 (0.699) | -4.40 (4.455)
  Cycle 2 | -0.95 (1.678) | -1.76 (3.427) | -1.17 (1.545) | -1.15 (1.556)
  Cycle 3: number analyzed (Participants) | 5 | 4 | 6 | 2
  Cycle 3 | 0.04 (1.076) | -1.00 (1.442) | -1.69 (1.429) | -3.90 (0.495)
  Cycle 4: number analyzed (Participants) | 5 | 4 | 6 | 2
  Cycle 4 | -0.51 (0.989) | -3.70 (3.252) | -2.54 (1.787) | -4.90 (0.495)

5. Secondary Outcome: Changes in the Mean Daily Numerical Rating Scale (NRS) Scores for the Worst Non-menstrual Pelvic Pain.
Description: as for outcome 3
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 2
score on a scale
  Cycle 1 | -0.09 (1.457) | -1.45 (0.926) | -0.61 (0.847) | -1.42 (0.693)
  Cycle 2: number analyzed (Participants) | 6 | 5 | 7 | 2
  Cycle 2 | -0.69 (1.484) | -2.71 (2.995) | -1.64 (1.354) | -1.22 (1.036)
  Cycle 3: number analyzed (Participants) | 5 | 5 | 6 | 2
  Cycle 3 | -0.77 (1.194) | -3.21 (3.390) | -1.39 (2.306) | -1.88 (2.632)
  Cycle 4: number analyzed (Participants) | 5 | 3 | 6 | 2
  Cycle 4 | -0.69 (1.236) | -2.04 (2.390) | -2.08 (1.274) | -3.37 (2.040)

6. Secondary Outcome: Changes in the Mean Daily Numerical Rating Scale (NRS) Scores for the Worst Dyspareunia on Days With Sexual Intercourse.
Description: as for outcome 3
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 3 | 6 | 1
score on a scale
  Cycle 1 | -1.62 (1.850) | -0.49 (1.088) | -1.69 (1.972) | -1.00 (NA) — Only 1 participant
  Cycle 2: number analyzed (Participants) | 5 | 3 | 4 | 0
  Cycle 2 | -1.43 (2.008) | -0.06 (0.756) | -1.50 (1.542) |
  Cycle 3: number analyzed (Participants) | 5 | 3 | 5 | 1
  Cycle 3 | -0.53 (1.514) | -0.29 (1.551) | -2.12 (2.791) | -7.00 (NA) — Only 1 participant
  Cycle 4: number analyzed (Participants) | 4 | 2 | 5 | 1
  Cycle 4 | -1.45 (1.468) | 0.85 (1.109) | -2.03 (0.864) | -5.00 (NA) — Only 1 participant

7. Secondary Outcome: Frequency of Avoiding Sexual Intercourse Due to Expected Pain
Description: The participants recorded daily if they had sexual intercourse, in an e-diary. For the days when participants did not have intercourse, the participant recorded if the reason for not having intercourse was because they expected pain: "Yes" (I did not have intercourse this day, because I expected pain) or "No" (I did not have intercourse this day, but this was not because I expected pain). The numbers represent the cumulative number of days with no intercourse, summed across all participants.
  In some cases, there are missing data as not every participant completed the e-diary for 100% of study days.
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Measure: Number; unit: Number of days
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 3
Number of days
  Baseline - Yes | 36 | 46 | 41 | 24
  Baseline - No | 103 | 94 | 154 | 48
  Cycle 1 - Yes | 38 | 20 | 35 | 22
  Cycle 1 - No | 116 | 107 | 158 | 28
  Cycle 2 - Yes | 34 | 13 | 29 | 11
  Cycle 2 - No | 107 | 109 | 153 | 40
  Cycle 3 - Yes | 30 | 23 | 31 | 1
  Cycle 3 - No | 112 | 106 | 122 | 51
  Cycle 4 - Yes | 29 | 11 | 28 | 3
  Cycle 4 - No | 94 | 67 | 117 | 64

8. Secondary Outcome: Changes in the Mean Daily Numerical Rating Scale (NRS) Scores for the Worst Impact of Endometriosis-related Pain on the Subject's Ability to Function.
Description: as for outcome 3
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 7 | 2
score on a scale
  Cycle 1 | -0.27 (1.095) | -1.45 (1.079) | -0.31 (0.741) | -1.77 (1.324)
  Cycle 2 | -0.53 (0.867) | -2.19 (3.194) | -0.95 (1.281) | -0.76 (1.518)
  Cycle 3: number analyzed (Participants) | 5 | 4 | 6 | 2
  Cycle 3 | -0.08 (1.438) | -1.44 (1.871) | -0.87 (1.847) | -2.02 (2.631)
  Cycle 4: number analyzed (Participants) | 5 | 3 | 6 | 2
  Cycle 4 | -0.32 (1.647) | -1.57 (2.203) | -1.48 (1.649) | -3.61 (1.678)

9. Secondary Outcome: Changes in the Mean Weekly Scores of the Endometriosis Health Profile-30 (EHP-30) Pain Impact Domain.
Description: Assessed weekly by participants in an e-Diary. EHP-30 is a quality-of-life questionnaire. Score ranges from 0-100 and lower score denotes improvement.
  Changes over 4 menstrual cycles.
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 2
score on a scale
  Cycle 1 | -5.54 (10.939) | -5.54 (11.787) | -7.03 (10.050) | -26.66 (18.146)
  Cycle 2: number analyzed (Participants) | 6 | 5 | 7 | 2
  Cycle 2 | -5.69 (16.059) | -13.53 (28.807) | -14.27 (8.470) | -4.12 (17.477)
  Cycle 3: number analyzed (Participants) | 6 | 5 | 6 | 2
  Cycle 3 | -3.19 (14.065) | -21.19 (31.336) | -13.70 (12.564) | -27.89 (27.253)
  Cycle 4: number analyzed (Participants) | 5 | 4 | 6 | 2
  Cycle 4 | -6.75 (15.743) | -24.75 (35.171) | -16.01 (8.624) | -31.68 (21.896)

10. Secondary Outcome: Changes in Vaginal Bleeding Pattern - Number of Days With Bleeding Related to Period
Description: The participants recorded daily if they had any vaginal bleeding during the past 24 hours, in an e-diary. Of the participants who had a bleeding, the participant recorded if this was menstrual bleeding: "Yes" (I had a vaginal bleeding that was menstrual bleeding) or "No" (I had a vaginal bleeding that was not menstrual bleeding). The numbers represent the cumulative number of days with vaginal bleeding, summed across all participants.
  In some cases, there are missing data as not every participant completed the e-diary for 100% of study days.
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Number; unit: Number of days
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 3
Number of days
  Bleeding related to period - Baseline Yes | 38 | 37 | 42 | 15
  Bleeding related to period - Baseline No | 11 | 0 | 10 | 2
  Bleeding related to period - Cycle 4 Yes | 29 | 16 | 33 | 17
  Bleeding related to period - Cycle 4 No | 3 | 5 | 2 | 0

11. Secondary Outcome: Changes in Vaginal Bleeding Pattern.
Description: The participants recorded daily if they had any vaginal bleeding during the past 24 hours, in an e-diary. Of the participants who had a bleeding, the participant recorded the assessed bleeding volume as either spotting (tiny amount of blood on underwear or panty liners), light bleeding (requiring 1-3 sanitary pads or tampons per day), moderate bleeding (requiring 4-6 sanitary pads or tampons per day), or heavy bleeding (requiring more than 6 sanitary pads or tampons per day). The numbers represent the cumulative number of days with vaginal bleeding, summed across all participants.
  In some cases, there are missing data as not every participant completed the e-diary for 100% of study days.
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Number; unit: Number of days
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 3
Number of days
  No bleeding - Baseline | 91 | 101 | 144 | 56
  Spotting - Baseline | 18 | 9 | 16 | 3
  Light - Baseline | 17 | 11 | 12 | 8
  Moderate - Baseline | 10 | 11 | 15 | 3
  Heavy - Baseline | 5 | 9 | 10 | 3
  No Bleeding - Cycle 4 | 91 | 57 | 110 | 50
  Spotting - Cycle 4 | 12 | 8 | 11 | 2
  Light - Cycle 4 | 8 | 7 | 9 | 9
  Moderate - Cycle 4 | 9 | 4 | 10 | 3
  Heavy - Cycle 4 | 3 | 2 | 5 | 3

12. Secondary Outcome: Percentage of Days With Mild and/or Strong Rescue Analgesics Used
Description: Assessed daily by participants in an e-Diary
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 7 | 2
percentage of days
  Cycle 1 - Any analgesics | 41.68 (31.961) | 26.04 (41.912) | 44.82 (35.052) | 3.57 (5.051)
  Cycle 1 - Mild analgesics | 41.68 (31.961) | 22.41 (43.522) | 44.82 (35.052) | 3.57 (5.051)
  Cycle 1 - Strong analgesics | 10.75 (22.649) | 5.12 (7.976) | 3.43 (9.071) | 0 (0)
  Cycle 2 - Any analgesics | 40.96 (37.699) | 25.33 (42.310) | 36.29 (39.131) | 20.37 (28.808)
  Cycle 2 - Mild analgesics | 40.96 (37.699) | 21.00 (44.215) | 36.29 (39.131) | 20.37 (28.808)
  Cycle 2 - Strong analgesics | 12.35 (30.241) | 10.99 (14.572) | 2.86 (7.559) | 0 (0)
  Cycle 3 - Any analgesics: number analyzed (Participants) | 5 | 4 | 6 | 2
  Cycle 3 - Any analgesics | 39.67 (40.008) | 32.25 (44.036) | 38.62 (44.213) | 13.46 (13.598)
  Cycle 3 - Mild analgesics: number analyzed (Participants) | 5 | 4 | 6 | 2
  Cycle 3 - Mild analgesics | 38.00 (36.920) | 29.47 (46.115) | 38.62 (44.213) | 13.46 (13.598)
  Cycle 3 - Strong analgesics: number analyzed (Participants) | 5 | 4 | 6 | 2
  Cycle 3 - Strong analgesics | 10.83 (24.224) | 10.13 (13.880) | 5.17 (12.670) | 0 (0)
  Cycle 4 - Any analgesics: number analyzed (Participants) | 5 | 3 | 6 | 2
  Cycle 4 - Any analgesics | 39.88 (35.135) | 5.93 (6.988) | 37.75 (44.143) | 2.56 (3.626)
  Cycle 4 - Mild analgesics: number analyzed (Participants) | 5 | 3 | 6 | 2
  Cycle 4 - Mild analgesics | 39.88 (35.135) | 1.39 (2.406) | 37.75 (44.143) | 2.56 (3.626)
  Cycle 4 - Strong analgesics: number analyzed (Participants) | 5 | 3 | 6 | 2
  Cycle 4 - Strong analgesics | 9.17 (20.497) | 4.55 (7.873) | 3.47 (8.505) | 0 (0)

13. Secondary Outcome: Total and Average Doses of Mild and/or Strong Rescue Analgesics Used
Description: Assessed daily by participants in an e-Diary
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 7 | 2
mg
  Total dose of mild analgesics - Cycle 1 | 8400.0 (7740.80) | 5680.0 (11389.12) | 14514.3 (14920.17) | 1200.0 (1697.06)
  Average dose of mild analgesics - Cycle 1 | 325.10 (339.854) | 213.27 (420.629) | 613.51 (665.765) | 42.86 (60.609)
  Total dose of mild analgesics - Cycle 2 | 11266.7 (15184.03) | 5480.0 (11594.48) | 13485.7 (17324.30) | 8600.0 (12162.24)
  Average dose of mild analgesics - Cycle 2 | 443.41 (557.172) | 230.28 (482.277) | 487.05 (613.429) | 318.52 (450.453)
  Total dose of mild analgesics - Cycle 3: number analyzed (Participants) | 5 | 4 | 6 | 2
  Total dose of mild analgesics - Cycle 3 | 10360.0 (11802.03) | 10650.0 (17070.34) | 16166.7 (17716.17) | 5500.0 (6646.80)
  Average dose of mild analgesics - Cycle 3: number analyzed (Participants) | 5 | 4 | 6 | 2
  Average dose of mild analgesics - Cycle 3 | 412.97 (490.864) | 333.19 (497.634) | 590.77 (648.496) | 211.54 (255.646)
  Total dose of mild analgesics - Cycle 4: number analyzed (Participants) | 5 | 3 | 6 | 2
  Total dose of mild analgesics - Cycle 4 | 9760.0 (11939.35) | 400.0 (692.82) | 15333.3 (21142.44) | 1200.0 (1697.06)
  Average dose of mild analgesics - Cycle 4: number analyzed (Participants) | 5 | 3 | 6 | 2
  Average dose of mild analgesics - Cycle 4 | 403.73 (507.562) | 16.00 (27.713) | 606.03 (824.589) | 30.77 (43.514)
  Total dose of strong analgesics - Cycle 1 | 1575.8 (3431.31) | 427.0 (668.22) | 697.1 (1844.47) | 0 (0)
  Average dose of strong analgesics - Cycle 1 | 66.93 (146.737) | 18.38 (30.108) | 27.89 (73.779) | 0 (0)
  Total dose of strong analgesics - Cycle 2 | 2541.7 (6225.79) | 854.0 (1086.93) | 915.0 (2420.86) | 0 (0)
  Average dose of strong analgesics - Cycle 2 | 94.42 (231.273) | 36.03 (45.793) | 30.50 (80.695) | 0 (0)
  Total dose of strong analgesics - Cycle 3: number analyzed (Participants) | 5 | 4 | 6 | 2
  Total dose of strong analgesics - Cycle 3 | 2013.0 (4501.20) | 1143.8 (1460.08) | 1575.8 (3859.99) | 0 (0)
  Average dose of strong analgesics - Cycle 3: number analyzed (Participants) | 5 | 4 | 6 | 2
  Average dose of strong analgesics - Cycle 3 | 79.38 (177.493) | 36.55 (44.327) | 54.34 (133.103) | 0 (0)
  Total dose of strong analgesics - Cycle 4: number analyzed (Participants) | 5 | 3 | 6 | 2
  Total dose of strong analgesics - Cycle 4 | 1159.0 (2591.60) | 305.0 (528.28) | 305.0 (747.09) | 0 (0)
  Average dose of strong analgesics - Cycle 4: number analyzed (Participants) | 5 | 3 | 6 | 2
  Average dose of strong analgesics - Cycle 4 | 46.14 (103.164) | 13.26 (22.968) | 12.71 (31.129) | 0 (0)

14. Secondary Outcome: Responder Rate
Description: Assessed as ≥30%, ≥50% and ≥70% reduction from the baseline in mean daily NRS score for the worst endometriosis-related pain, dysmenorrhea and non-menstrual pelvic pain and for the worst endometriosis-related pain impact
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 4 | 6 | 2
percentage of participants
  ≥30% reduction - endometriosis-related pain | 20.0 | 50.0 | 33.3 | 100
  ≥30% reduction - dysmenorrhea | 0 | 75.0 | 50.0 | 100
  ≥30% reduction - non-menstrual pelvic pain | 20.0 | 50.0 | 33.3 | 100
  ≥30% reduction - impact on the subject's ability to function | 20.0 | 50.0 | 33.3 | 100
  ≥50% reduction - endometriosis-related pain | 0 | 25.0 | 33.3 | 50.0
  ≥50% reduction - dysmenorrhea | 0 | 50.0 | 33.3 | 100
  ≥50% reduction - non-menstrual pelvic pain | 20.0 | 25.0 | 33.3 | 50.0
  ≥50% reduction - impact on the subject's ability to function | 0 | 50.0 | 33.3 | 50.0
  ≥70% reduction - endometriosis-related pain | 0 | 0 | 16.7 | 0
  ≥70% reduction - dysmenorrhea | 0 | 25.0 | 16.7 | 0
  ≥70% reduction - non-menstrual pelvic pain | 0 | 25.0 | 16.7 | 0
  ≥70% reduction - impact on the subject's ability to function | 0 | 25.0 | 16.7 | 0

15. Secondary Outcome: Changes in the Mean Individual and Total Symptom and Sign Severity Scores
Description: Assessed by the Biberoglu and Behrman (B&B) scale which is a 4-point scale with 0=none and 3=severe.
  The scores are the mean individual scores.
  The B&B scale consists of two parts. The first part of the B&B scale evaluates symptoms of endometriosis (i.e. pain). There are 3 subscales: pelvic pain(A, 0=none and 3=severe), dysmenorrhea (B, 0=none and 3=severe), and dyspareunia(C, 0=none and 3=severe). The total pelvic pain score is the sum of the three scores, i.e. A+B+C, which can range from 0 to 9. The second part of the B&B scale evaluates signs of endometriosis. There are 2 subscales pelvic tenderness (D, 0=none and 3=severe) and induration (E, 0=none and 3=severe) based on findings from a pelvic examination. The total physical pain score is the sum of the two scores, i.e. D+E, which can range from 0 to 6. The total symptom and sign severity score is the sum of all five scores, i.e. A+B+C+D+E, which can range from 0 to 15.
  The values are the change from baseline to cycle 4.
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
score on a scale
  Total pelvic pain score | -1.0 (1.73) | -3.0 (5.66) | -2.4 (2.51) | -5.0 (NA) — Only 1 participant
  Total physical sign pain score | -1.7 (1.53) | -1.5 (0.71) | -2.2 (1.48) | -1.0 (NA) — Only 1 participant
  Total symptom and sign severity score | -2.7 (3.21) | -4.5 (4.95) | -4.6 (3.91) | -6.0 (NA) — Only 1 participant

16. Secondary Outcome: Changes in the Endometriosis Health Profile-30 (EHP-30) Scores
Description: Assessed by the EHP-30 quality-of-life questionnaire completed by participants. Score ranges from 0-100 with lower score denoting improvement.
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 5 | 8 | 2
score on a scale
  Cycle 1 | -7.2 (15.22) | -12.8 (18.09) | -8.8 (13.86) | -39.5 (74.25)
  Cycle 2: number analyzed (Participants) | 5 | 5 | 7 | 2
  Cycle 2 | -2.0 (22.55) | -12.0 (25.88) | -19.7 (15.52) | -49.5 (68.59)
  Cycle 3: number analyzed (Participants) | 4 | 5 | 6 | 2
  Cycle 3 | -2.8 (20.98) | -12.4 (26.02) | -18.7 (15.25) | -14.0 (11.31)
  Cycle 4: number analyzed (Participants) | 4 | 4 | 6 | 2
  Cycle 4 | -4.0 (33.79) | -23.3 (25.63) | -23.3 (12.86) | -50.5 (31.82)

17. Secondary Outcome: Changes in Patient Global Impression of Severity (PGIS) Scores
Description: Assessed by the PGIS scale completed by participants. PGIS is a 6-point scale depicting a participant's rating of their current conditions from "good" to "bad".
  It ranges from 0 (none) to 5 (very severe).
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 4 | 6 | 2
Participants
  Endometriosis-related pain during the last menstrual cycle: No Change | 2 | 1 | 3 | 0
  Endometriosis-related pain during the last menstrual cycle: Decreased score | 2 | 3 | 3 | 2
  Endometriosis-related pain during the last menstrual cycle: Increased score | 0 | 0 | 0 | 0
  Endometriosis-related pain during the menstrual bleeding days of the last menstrual cycle: No Change | 2 | 0 | 1 | 0
  Endometriosis-related pain during the menstrual bleeding days of the last menstrual cycle: Decreased score | 2 | 4 | 4 | 2
  Endometriosis-related pain during the menstrual bleeding days of the last menstrual cycle: Increased score | 0 | 0 | 1 | 0
  Endometriosis-related pain during non-menstrual bleeding days of the last menstrual cycle: No Change | 1 | 0 | 2 | 0
  Endometriosis-related pain during non-menstrual bleeding days of the last menstrual cycle: Decreased score | 2 | 4 | 4 | 2
  Endometriosis-related pain during non-menstrual bleeding days of the last menstrual cycle: Increased score | 1 | 0 | 0 | 0
  Impact of endometriosis-related pain on daily activities during the last menstrual cycle: No Change | 2 | 0 | 0 | 0
  Impact of endometriosis-related pain on daily activities during the last menstrual cycle: Decreased score | 2 | 4 | 5 | 2
  Impact of endometriosis-related pain on daily activities during the last menstrual cycle: Increased score | 0 | 0 | 1 | 0
  Impact of pain on daily activities during the menstrual bleeding days of the last menstrual cycle: No Change | 1 | 0 | 1 | 0
  Impact of pain on daily activities during the menstrual bleeding days of the last menstrual cycle: Decreased score | 3 | 4 | 5 | 2
  Impact of pain on daily activities during the menstrual bleeding days of the last menstrual cycle: Increased score | 0 | 0 | 0 | 0
  Impact of pain on daily activities during non-menstrual bleeding days of the last menstrual cycle: No Change | 1 | 1 | 1 | 0
  Impact of pain on daily activities during non-menstrual bleeding days of the last menstrual cycle: Decreased score | 3 | 3 | 4 | 2
  Impact of pain on daily activities during non-menstrual bleeding days of the last menstrual cycle: Increased score | 0 | 0 | 1 | 0

18. Secondary Outcome: Patient Global Impression of Change (PGIC) Scores
Description: Assessed by the PGIC scale completed by participants. PGIC is a 7-point scale depicting a patient's rating of their overall improvement from "good" to "bad".
Time Frame: At cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 4 | 6 | 2
Participants
  Change in endometriosis-related pain: Very much improved | 0 | 1 | 0 | 2
  Change in endometriosis-related pain: Much improved | 1 | 1 | 2 | 0
  Change in endometriosis-related pain: Minimally improved | 3 | 2 | 4 | 0
  Change in endometriosis-related pain: No change | 1 | 0 | 0 | 0
  Change in endometriosis-related pain: Very much worse | 0 | 0 | 0 | 0
  Change in dysmenorrhea: Very much improved | 0 | 1 | 0 | 2
  Change in dysmenorrhea: Much improved | 0 | 1 | 2 | 0
  Change in dysmenorrhea: Minimally improved | 5 | 1 | 2 | 0
  Change in dysmenorrhea: No change | 0 | 1 | 1 | 0
  Change in dysmenorrhea: Very much worse | 0 | 0 | 1 | 0
  Change of non-menstrual pelvic pain: Very much improved | 1 | 1 | 0 | 1
  Change of non-menstrual pelvic pain: Much improved | 0 | 1 | 2 | 0
  Change of non-menstrual pelvic pain: Minimally improved | 3 | 2 | 3 | 0
  Change of non-menstrual pelvic pain: No change | 1 | 0 | 1 | 1
  Change of non-menstrual pelvic pain: Very much worse | 0 | 0 | 0 | 0
  Change in the overall impact of endometriosis-related pain on daily activities: Very much improved | 0 | 1 | 0 | 2
  Change in the overall impact of endometriosis-related pain on daily activities: Much improved | 0 | 1 | 2 | 0
  Change in the overall impact of endometriosis-related pain on daily activities: Minimally improved | 4 | 1 | 3 | 0
  Change in the overall impact of endometriosis-related pain on daily activities: No change | 1 | 1 | 1 | 0
  Change in the overall impact of endometriosis-related pain on daily activities: Very much worse | 0 | 0 | 0 | 0
  Change in endometriosis-related pain impact during their menstrual periods: Very much improved | 0 | 1 | 0 | 2
  Change in endometriosis-related pain impact during their menstrual periods: Much improved | 0 | 0 | 2 | 0
  Change in endometriosis-related pain impact during their menstrual periods: Minimally improved | 4 | 1 | 3 | 0
  Change in endometriosis-related pain impact during their menstrual periods: No change | 1 | 2 | 0 | 0
  Change in endometriosis-related pain impact during their menstrual periods: Very much worse | 0 | 0 | 1 | 0
  Change in the endometriosis related pain impact during non-menstrual periods: Very much improved | 0 | 1 | 0 | 2
  Change in the endometriosis related pain impact during non-menstrual periods: Much improved | 2 | 1 | 2 | 0
  Change in the endometriosis related pain impact during non-menstrual periods: Minimally improved | 2 | 1 | 3 | 0
  Change in the endometriosis related pain impact during non-menstrual periods: No change | 1 | 1 | 0 | 0
  Change in the endometriosis related pain impact during non-menstrual periods: Very much worse | 0 | 0 | 1 | 0

19. Secondary Outcome: Plasma Concentration of Quinagolide and Metabolites
Description: Assessed by blood samples collection
Time Frame: Within 5 days after first ring insertion and at around 1 month, 3 months, 3.5 months and 4 months after baseline (each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg
Number analyzed (Participants) | 6 | 4 | 7
pg/mL
  Within 1-5 days of first ring inserting | 3.04 (1.09) | 7.77 (3.94) | 10.5 (8.79)
  Luteinizing hormone surge + 7 days visit during cycle 1: number analyzed (Participants) | 3 | 2 | 6
  Luteinizing hormone surge + 7 days visit during cycle 1 | 1.84 (1.31) | 2.36 (0.750) | 7.10 (2.36)
  Return of Menses + 7 days visit during cycle 1: number analyzed (Participants) | 5 | 3 | 6
  Return of Menses + 7 days visit during cycle 1 | 1.22 (0.632) | 1.52 (0.54) | 3.22 (1.70)
  Return of Menses+7 days visit during cycle 3: number analyzed (Participants) | 4 | 4 | 5
  Return of Menses+7 days visit during cycle 3 | 1.44 (0.578) | 2.00 (0.98) | 5.70 (5.55)
  Luteinizing hormone surge + 7 days visit during cycle 4: number analyzed (Participants) | 5 | 1 | 5
  Luteinizing hormone surge + 7 days visit during cycle 4 | 2.08 (0.65) | 2.92 (NA) — Only 1 participant | 5.13 (2.91)
  Return of Menses+7 days visit during cycle 4: number analyzed (Participants) | 5 | 3 | 5
  Return of Menses+7 days visit during cycle 4 | 1.47 (0.799) | 2.07 (0.85) | 3.41 (2.43)

20. Secondary Outcome: Serum Levels of Mid-luteal Phase Progesterone
Description: Assessed by blood samples collection
Time Frame: At baseline and cycle 4 (around 3.5 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 3
ng/mL
  Baseline | 8.29 (4.984) | 8.49 (6.343) | 7.04 (6.014) | 8.57 (1.537)
  Cycle 4: number analyzed (Participants) | 5 | 2 | 5 | 2
  Cycle 4 | 9.55 (7.389) | 6.00 (6.505) | 6.56 (6.382) | 0.05 (0.000)

21. Secondary Outcome: Number of Subjects With Serum Mid-luteal Progesterone Levels ≥25 Nmol/L (7.9 ng/ml)
Description: Assessed by blood samples collection
Time Frame: At baseline and cycle 4 (around 3.5 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 3
Participants
  Baseline: < 7.9 | 2 | 2 | 4 | 1
  Baseline: >= 7.9 | 4 | 3 | 4 | 2
  Cycle 4: number analyzed (Participants) | 5 | 2 | 5 | 2
  Cycle 4: < 7.9 | 3 | 1 | 2 | 2
  Cycle 4: >= 7.9 | 2 | 1 | 3 | 0

22. Secondary Outcome: Serum Levels of Estradiol
Description: Assessed by blood samples collection
Time Frame: At baseline and cycle 4 (around 3.5 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 7 | 3
pmol/L
  Baseline | 328.2 (105.46) | 534.4 (215.68) | 350.0 (141.05) | 431.6 (67.41)
  Cycle 4: number analyzed (Participants) | 5 | 2 | 5 | 2
  Cycle 4 | 415.6 (84.52) | 278.8 (229.21) | 552.3 (267.16) | 142.8 (10.90)

23. Secondary Outcome: Serum Levels of Prolactin
Description: Assessed by blood samples collection
Time Frame: At baseline and cycle 4 (around 3.5 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 3
ng/mL
  Baseline | 8.0 (2.40) | 13.2 (8.25) | 10.0 (2.95) | 13.4 (0.69)
  Cycle 4: number analyzed (Participants) | 5 | 2 | 5 | 2
  Cycle 4 | 10.7 (5.04) | 11.3 (2.97) | 9.0 (2.50) | 35.7 (20.22)

24. Secondary Outcome: Serum Levels of Thyrotropin (TSH)
Description: Assessed by blood samples collection
Time Frame: At baseline and cycle 4 (around 3.5 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 5 | 8 | 3
uIU/mL
  Baseline | 1.9 (0.97) | 2.1 (1.25) | 1.3 (0.56) | 2.7 (2.14)
  Cycle 4: number analyzed (Participants) | 5 | 2 | 5 | 1
  Cycle 4 | 1.7 (0.55) | 2.1 (1.17) | 1.2 (0.78) | 2.3 (NA) — Only 1 participant

25. Secondary Outcome: Serum Levels of Insulin-like Growth Factor-1 (IGF-1)
Description: Assessed by blood samples collection
Time Frame: At baseline and cycle 4 (around 3.5 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 7 | 3
ng/mL
  Baseline | 216.7 (50.11) | 221.1 (89.37) | 166.2 (59.58) | 188.7 (12.57)
  Cycle 4: number analyzed (Participants) | 5 | 2 | 5 | 2
  Cycle 4 | 211.5 (38.37) | 208.3 (142.27) | 158.1 (53.32) | 169.9 (12.73)

26. Secondary Outcome: Changes in Bone Turnover Markers, Determined by Bone Resorption Marker Serum C-terminal Crosslinking Telopeptide of Type 1 Collagen (s-CTx)
Description: Assessed by blood samples collection. Changes from baseline to cycle 4
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 2 | 5 | 2
ng/mL | -0.060 (0.1210) | 0.277 (0.3026) | 0.067 (0.0685) | -0.031 (0.0354)

27. Secondary Outcome: Changes in Bone Turnover Markers, Determined by Bone Formation Marker Serum Procollagen Type I N Propeptide (s-PINP)
Description: Assessed by blood samples collection. Changes from baseline to cycle 4
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 2 | 4 | 1
ng/mL | -1.4 (9.56) | -3.5 (6.36) | 10.3 (20.12) | -21.0 (NA) — Only 1 participant

28. Secondary Outcome: Changes in ECG Parameters Including PR Interval at Cycle 4
Description: Assessed by 12-lead ECG
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 4 | 5 | 2
msec | -1.8 (11.17) | 8.0 (8.72) | 1.0 (11.66) | -2.5 (2.12)

29. Secondary Outcome: Changes in ECG Parameters Including QRS Duration at Cycle 4
Description: Assessed by 12-lead ECG
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 4 | 5 | 2
msec | -0.2 (4.82) | 5.0 (5.83) | 2.8 (7.19) | -7.5 (9.19)

30. Secondary Outcome: Changes in ECG Parameters Including QT Interval at Cycle 4
Description: Assessed by 12-lead ECG
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 4 | 5 | 2
msec | -1.2 (22.33) | -7.5 (23.61) | 18.0 (30.32) | 7.0 (5.66)

31. Secondary Outcome: Changes in ECG Parameters Including QTcF Interval at Cycle 4
Description: Assessed by 12-lead ECG
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 5 | 4 | 5 | 2
msec | -6.2 (6.18) | 1.5 (11.39) | 3.2 (13.22) | -17.5 (33.23)

32. Secondary Outcome: Proportion of Subjects With Abnormal Clinically Significant Echocardiography Findings Indicating Valvular Heart Disease
Description: Assessed by echocardiography.
  Each echocardiography was to be assessed as normal or abnormal according to American College of Cardiology/American Heart Association guidelines for valvular heart disease. If abnormal, the level of valvular regurgitation and valvular stenosis was specified as mild, moderate or severe and valvular structure was evaluated as well.
  Measured at cycle 4.
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 3
Participants | 0 | 0 | 0 | 0

33. Secondary Outcome: Proportion of Subjects Identified With Potential Impulse Control Disorders
Description: Assessed by the questionnaire for impulsive-compulsive disorders completed by participants.
  Measured at cycle 4.
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 8 | 2
Participants | 1 | 0 | 0 | 0

34. Secondary Outcome: Frequency and Intensity of Adverse Events
Description: Assessed by an Adverse Events Log completed by the Investigator
Time Frame: From signing informed consent through study completion, around 8 months
Measure: Number; unit: participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 3
participants
  Treatment emergent adverse events | 4 | 3 | 5 | 2
  Mild adverse events | 4 | 2 | 4 | 2
  Moderate adverse events | 2 | 2 | 2 | 2
  Severe adverse events | 0 | 1 | 0 | 0

35. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Albumin
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
g/L | -0.5 (3.00) | 0.5 (2.12) | -2.8 (2.28) | -3.0 (NA) — Only 1 participant

36. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Alkaline Phosphatase
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
IU/L | -16.5 (20.94) | 26.5 (45.96) | -7.2 (14.62) | -13.0 (NA) — Only 1 participant

37. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Alanine Aminotransferase
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
IU/L | -8.3 (23.26) | 46.0 (69.30) | -5.8 (6.38) | -3.0 (NA) — Only 1 participant

38. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Aspartate Aminotransferase
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
IU/L | -5.3 (14.57) | 26.5 (41.72) | -0.6 (1.14) | 4.0 (NA) — Only 1 participant

39. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Bicarbonate
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
mmol/L | -0.8 (2.63) | 0.5 (3.54) | -0.2 (1.92) | -2.0 (NA) — Only 1 participant

40. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Direct Bilirubin
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
umol/L | 0.0 (0.0) | 0.0 (0.0) | -0.7 (0.72) | 0.0 (0.0)

41. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Bilirubin
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
umol/L | 1.3 (2.57) | 4.3 (3.63) | -2.1 (2.23) | 1.7 (NA) — Only 1 participant

42. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Calcium
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
mmol/L | 0.0 (0.06) | 0.0 (0.05) | -0.1 (0.07) | -0.1 (NA) — Only 1 participant

43. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Cholesterol
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
mmol/L | 0.7 (0.46) | 0.5 (0.49) | 0.1 (0.27) | -0.1 (NA) — Only 1 participant

44. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Chloride
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 2
mmol/L | 0.8 (1.71) | 1.0 (0.00) | 1.4 (2.51) | 2.5 (2.12)

45. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Creatinine
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
umol/L | -3.3 (13.39) | -10.6 (3.75) | 0.0 (7.26) | 0.9 (NA) — Only 1 participant

46. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Gamma Glutamyl Transferase
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
IU/L | -3.5 (9.75) | 11.0 (14.14) | -2.8 (11.32) | -9.0 (NA) — Only 1 participant

47. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Glucose
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
mmol/L | -0.3 (0.40) | -0.6 (0.59) | -0.1 (0.49) | 4.8 (NA) — Only 1 participant

48. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Potassium
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 2
mmol/L | -0.2 (0.58) | -0.1 (0.00) | -0.3 (0.32) | -0.5 (0.00)

49. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Lactate Dehydrogenase
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
IU/L | -11.8 (14.86) | 35.0 (55.15) | -16.0 (14.68) | 8.0 (NA) — Only 1 participant

50. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Phosphate
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
mmol/L | 0.1 (0.08) | -0.1 (0.43) | 0.0 (0.12) | 0.0 (NA) — Only 1 participant

51. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Protein
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
g/L | -0.8 (4.35) | 0.0 (2.83) | -3.4 (3.65) | -5.0 (NA) — Only 1 participant

52. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Sodium
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 2
mmol/L | 1.5 (1.73) | -1.5 (3.54) | 1.2 (2.39) | 0.5 (4.95)

53. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Urate
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
umol/L | -5.9 (31.85) | -23.8 (50.47) | 10.7 (64.80) | 41.6 (NA) — Only 1 participant

54. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters: Urea Nitrogen
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
mmol/L | 0.3 (2.21) | -2.0 (0.76) | -0.4 (0.84) | -0.7 (NA) — Only 1 participant

55. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Basophils Absolute
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Basophils Absolute (%)
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
Basophils Absolute (%) | -0.3 (0.25) | -0.4 (0.21) | 0.0 (0.05) | 0.1 (NA) — Only 1 participant

56. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Basophils
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: *10^3 cells/uL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
*10^3 cells/uL | 0.0 (0.03) | 0.0 (0.02) | 0.0 (0.02) | 0.0 (NA) — Only 1 participant

57. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Eosinophils Absolute
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Eosinophils Absolute (%)
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
Eosinophils Absolute (%) | -0.6 (0.71) | -0.3 (2.19) | -1.4 (3.73) | 0.0 (NA) — Only 1 participant

58. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Eosinophils
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: *10^3 cells/uL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
*10^3 cells/uL | -0.1 (0.02) | -0.1 (0.14) | 0.0 (0.13) | 0.0 (NA) — Only 1 participant

59. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Hematocrit
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: RATIO
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
RATIO | 0.0 (0.03) | 0.0 (0.02) | 0.0 (0.03) | 0.0 (NA) — Only 1 participant

60. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Hemoglobin
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
g/L | 1.3 (10.07) | -1.5 (14.85) | -6.0 (7.87) | 0.0 (NA) — Only 1 participant

61. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Lymphocytes Absolute
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lymphocytes Absolute (%)
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
Lymphocytes Absolute (%) | 2.5 (1.96) | -0.6 (0.35) | -2.1 (8.22) | 3.9 (NA) — Only 1 participant

62. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Lymphocytes
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: *10^3 cells/uL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
*10^3 cells/uL | 0.3 (0.39) | -0.2 (0.54) | -0.1 (0.43) | 0.3 (NA) — Only 1 participant

63. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Ery. Mean Corpuscular Hemoglobin
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/cell
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
pg/cell | 0.3 (0.58) | 0.0 (0.0) | -0.2 (0.45) | 0.0 (NA) — Only 1 participant

64. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Ery. Mean Corpuscular HGB Concentration
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
mmol/L | 0.2 (0.72) | 0.3 (1.32) | -0.1 (0.52) | 1.2 (NA) — Only 1 participant

65. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Ery. Mean Corpuscular Volume
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
fL | 0.0 (2.65) | 0.5 (3.54) | 0.2 (1.64) | -3.0 (NA) — Only 1 participant

66. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Monocytes Absolute
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Monocytes Absolute (%)
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
Monocytes Absolute (%) | -2.1 (0.26) | -2.2 (1.34) | -0.1 (1.32) | 0.6 (NA) — Only 1 participant

67. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Monocytes
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: *10^3 cells/uL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
*10^3 cells/uL | -0.2 (0.03) | -0.2 (0.04) | 0.0 (0.13) | 0.0 (NA) — Only 1 participant

68. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Neutrophils Absolute
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Neutrophils Absolute (%)
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
Neutrophils Absolute (%) | 0.6 (2.74) | 3.4 (2.90) | 3.7 (7.28) | -4.6 (NA) — Only 1 participant

69. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Neutrophils
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: *10^3 cells/uL
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
*10^3 cells/uL | 0.3 (1.37) | 0.0 (1.67) | 0.1 (1.52) | -0.3 (NA) — Only 1 participant

70. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Platelets
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
10^9 cells/L | -10.3 (26.54) | 36.5 (50.20) | 1.8 (33.33) | 12.0 (NA) — Only 1 participant

71. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Erythrocytes
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
10^12 cells/L | -0.1 (0.35) | -0.1 (0.42) | -0.2 (0.24) | -0.1 (NA) — Only 1 participant

72. Secondary Outcome: Changes in Circulating Levels of Clinical Haematology Parameters: Leukocytes
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 3 | 2 | 5 | 1
10^9 cells/L | 0.3 (1.72) | -0.5 (2.05) | 0.0 (1.63) | 0.0 (NA) — Only 1 participant

73. Secondary Outcome: Urinalysis Parameters (Protein, Glucose, Bilirubin, pH, Nitrite, Ketone, Urobilinogen, Blood, Leukocytes, and Specific Gravity)
Description: Assessed by urine sample collection (dip-stick test). Overall Urinalysis Result.
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 1 | 1 | 2 | 2
Participants
  Normal overall urinalysis result | 1 | 1 | 2 | 2
  Abnormal overall urinalysis result | 0 | 0 | 0 | 0

74. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Changes in Circulating Levels of Clinical Chemistry Parameters
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
Participants | 0 | 0 | 0 | 0

75. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Changes in Circulating Levels of Clinical Haematology Parameters
Description: Assessed by blood samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 4 | 2 | 5 | 1
Participants | 0 | 0 | 0 | 0

76. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Changes in Urinalysis Parameters
Description: Assessed by urine samples collection
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 1 | 1 | 2 | 2
Participants | 0 | 0 | 0 | 0

77. Secondary Outcome: Frequency and Intensity of Ring Acceptability Parameters: Insertion of the Vaginal Ring
Description: Assessed by a questionnaire completed by participants, addressing ring insertion
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 7 | 2
Participants
  Cycle 1: Easy | 2 | 3 | 6 | 2
  Cycle 1: Easier than the previous ring | 3 | 2 | 0 | 0
  Cycle 1: Difficult | 1 | 0 | 0 | 0
  Cycle 1: Not Applicable (I was not given a new ring) | 0 | 0 | 1 | 0
  Cycle 2: Easy | 5 | 4 | 7 | 2
  Cycle 2: Easier than the previous ring | 1 | 1 | 0 | 0
  Cycle 2: Difficult | 0 | 0 | 0 | 0
  Cycle 2: Not Applicable (I was not given a new ring) | 0 | 0 | 0 | 0
  Cycle 3: number analyzed (Participants) | 4 | 4 | 6 | 2
  Cycle 3: Easy | 3 | 4 | 5 | 2
  Cycle 3: Easier than the previous ring | 1 | 0 | 1 | 0
  Cycle 3: Difficult | 0 | 0 | 0 | 0
  Cycle 3: Not Applicable (I was not given a new ring) | 0 | 0 | 0 | 0
  Cycle 4: number analyzed (Participants) | 3 | 3 | 5 | 1
  Cycle 4: Easy | 1 | 2 | 4 | 1
  Cycle 4: Easier than the previous ring | 0 | 0 | 1 | 0
  Cycle 4: Difficult | 0 | 0 | 0 | 0
  Cycle 4: Not Applicable (I was not given a new ring) | 2 | 1 | 0 | 0

78. Secondary Outcome: Frequency and Intensity of Ring Acceptability Parameters: Removal of the Vaginal Ring
Description: Assessed by a questionnaire completed by participants, addressing ring removal.
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 7 | 2
Participants
  Cycle 1: Easy | 6 | 5 | 6 | 2
  Cycle 1: Difficult | 0 | 0 | 1 | 0
  Cycle 2: Easy | 6 | 5 | 7 | 1
  Cycle 2: Difficult | 0 | 0 | 0 | 1
  Cycle 3: number analyzed (Participants) | 4 | 4 | 6 | 2
  Cycle 3: Easy | 4 | 4 | 6 | 2
  Cycle 3: Difficult | 0 | 0 | 0 | 0
  Cycle 4: number analyzed (Participants) | 3 | 3 | 5 | 1
  Cycle 4: Easy | 3 | 3 | 5 | 1
  Cycle 4: Difficult | 0 | 0 | 0 | 0

79. Secondary Outcome: Frequency and Intensity of Ring Acceptability Parameters: Felt the Ring
Description: Assessed by a questionnaire completed by participants, addressing any feeling of the ring while the ring is in the body.
Time Frame: From baseline to menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Quinagolide 360 µg | Quinagolide 720 µg | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 6 | 5 | 7 | 2
Participants
  Cycle 1: Never | 0 | 1 | 3 | 1
  Cycle 1: Occasionally | 6 | 2 | 4 | 0
  Cycle 1: Frequently | 0 | 2 | 0 | 0
  Cycle 1: Always | 0 | 0 | 0 | 1
  Cycle 2: Never | 0 | 2 | 2 | 1
  Cycle 2: Occasionally | 5 | 3 | 4 | 1
  Cycle 2: Frequently | 1 | 0 | 0 | 0
  Cycle 2: Always | 0 | 0 | 1 | 0
  Cycle 3: number analyzed (Participants) | 4 | 4 | 6 | 2
  Cycle 3: Never | 1 | 1 | 2 | 1
  Cycle 3: Occasionally | 2 | 3 | 3 | 1
  Cycle 3: Frequently | 1 | 0 | 0 | 0
  Cycle 3: Always | 0 | 0 | 1 | 0
  Cycle 4: number analyzed (Participants) | 3 | 3 | 5 | 1
  Cycle 4: Never | 1 | 0 | 1 | 1
  Cycle 4: Occasionally | 2 | 3 | 3 | 0
  Cycle 4: Frequently | 0 | 0 | 0 | 0
  Cycle 4: Always | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from signing of the informed consent until end-of-trial (around 8 months).
Description: Adverse events were recorded from signing of the informed consent until end-of-trial (around 8 months). All AEs occurring after start of first administration of IMP and before the follow-up visit were considered treatment-emergent.
Groups:
- Quinagolide 360 µg - Part A: Vaginal ring containing Quinagolide 360 μg, with daily target release rate of 4.5 μg
  Quinagolide 360 µg: Vaginal ring containing quinagolide 360 µg for daily releases
  Part A is cycle 1-4.
- Quinagolide 720 µg - Part A: Vaginal ring containing Quinagolide 720 μg, with daily target release rate of 9 μg
  Quinagolide 720 µg: Vaginal ring containing quinagolide 720 µg for daily releases.
  Part A is cycle 1-4.
- Quinagolide 1080 µg - Part A: Vaginal ring containing Quinagolide 1080 μg, with daily target release rate of 13.5 μg
  Quinagolide 1080 µg: Vaginal ring containing quinagolide 1080 µg for daily releases.
  Part A is cycle 1-4.
- Placebo - Part A: Vaginal ring containing matching placebo
  Placebo: Matching placebo.
  Only Part A. No participants were exposed to placebo vaginal ring during Part B of the trial.
- Quinagolide 360 µg - Part B: Vaginal ring containing Quinagolide 360 μg, with daily target release rate of 4.5 μg
  Quinagolide 360 µg: Vaginal ring containing quinagolide 360 µg for daily releases
  Part B is cycle 5-8.
- Quinagolide 720 µg - Part B: Vaginal ring containing Quinagolide 720 μg, with daily target release rate of 9 μg
  Quinagolide 720 µg: Vaginal ring containing quinagolide 720 µg for daily releases.
  Part B is cycle 5-8.
  2 participants received Quinagolide 720 µg for both Part A and Part B (8 cycles total) and 1 participant received placebo for Part A (4 cycles) and Quinagolide 720 µg for Part B (4 cycles).
- Quinagolide 1080 µg - Part B: Vaginal ring containing Quinagolide 1080 μg, with daily target release rate of 13.5 μg
  Quinagolide 1080 µg: Vaginal ring containing quinagolide 1080 µg for daily releases.
  Part B is cycle 5-8.
  6 participants received Quinagolide 1080 µg for both Part A and Part B (8 cycles total) and 1 participant received placebo for Part A (4 cycles) and Quinagolide 1080 µg for Part B (4 cycles).
Arm/Group | Quinagolide 360 µg - Part A | Quinagolide 720 µg - Part A | Quinagolide 1080 µg - Part A | Placebo - Part A | Quinagolide 360 µg - Part B | Quinagolide 720 µg - Part B | Quinagolide 1080 µg - Part B
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/8 | 0/3 | 0/3 | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/8 | 0/3 | 0/3 | 0/3 | 0/7
Other Adverse Events (participants affected / at risk) | 4/6 | 3/5 | 2/8 | 2/3 | 1/3 | 2/3 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinagolide 360 µg - Part A (N=6) | Quinagolide 720 µg - Part A (N=5) | Quinagolide 1080 µg - Part A (N=8) | Placebo - Part A (N=3) | Quinagolide 360 µg - Part B (N=3) | Quinagolide 720 µg - Part B (N=3) | Quinagolide 1080 µg - Part B (N=7)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
obsessive-compulsive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial vaginosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Uterine disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT03692403/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT03692403/SAP_001.pdf